CLINICAL TRIAL: NCT02348593
Title: A Twelve-week, Double-blind, Placebo-controlled, Randomized, Parallel-group, Multicenter Study of the Safety and Efficacy of JZP-110 [(R)-2-amino-3-phenylpropylcarbamate Hydrochloride] in the Treatment of Excessive Sleepiness in Subjects With Narcolepsy
Brief Title: "Twelve-week Study of the Safety and Efficacy of JZP-110 in the Treatment of Excessive Sleepiness in Narcolepsy"
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-002
Record Dates: First submitted 2015-01-15; First posted 2015-01-28 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 75 mg of JZP-110 (Active Comparator): Once Daily Dosing
  Interventions: Drug: JZP-110
- 150 mg JZP-110 (Active Comparator): Once Daily Dosing
  Interventions: Drug: JZP-110
- 300 mg of JZP-110 (Active Comparator): Once Daily Dosing
  Interventions: Drug: JZP-110
- Placebo (Placebo Comparator): Once Daily Dosing
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: JZP-110
  Arms: 150 mg JZP-110; 300 mg of JZP-110; 75 mg of JZP-110
Drug: Placebo oral tablet
  Arms: Placebo

SUMMARY:
This trial is a 12-week, randomized, double-blind, placebo controlled, multicenter, 4-treatment parallel group study of the safety and efficacy of JZP-110 in the treatment of excessive sleepiness in adult subjects with narcolepsy.

ELIGIBILITY:
Major Inclusion Criteria:

1. Males and females between 18 and 75 years of age, inclusive
2. Diagnosis of narcolepsy according to ICSD-3 or DSM-5 criteria
3. Body mass index from 18 to <45 kg/m2
4. Consent to use a medically acceptable method of contraception
5. Willing and able to provide written informed consent

Major Exclusion Criteria:

1. Female subjects who are pregnant, nursing, or lactating
2. Moderate or severe sleep apnea on the baseline PSG.
3. Any other clinically relevant medical, behavioral, or psychiatric disorder other than narcolepsy that is associated with excessive sleepiness
4. History or presence of bipolar disorder, bipolar related disorders, schizophrenia, schizophrenia spectrum disorders, or other psychotic disorders according to DSM-5 criteria
5. History or presence of any acutely unstable medical condition, behavioral or psychiatric disorder (including active suicidal ideation), or surgical history that could affect the safety of the subject or interfere with study efficacy, safety, PK assessments, or the ability of the subject to complete the trial per the judgment of the Investigator
6. History of bariatric surgery within the past year or a history of any gastic bypass procedure
7. Presence or history of significant cardiovascular disease
8. Use of any over-the-counter (OTC) or prescription medications that could affect the evaluation of excessive sleepiness
9. Use of any medications that could affect the evaluation of cataplexy
10. Received an investigational drug in the past 30 days or five half-lives (whichever is longer)
11. Previous exposure to or participation in a previous clinical trial of JZP-110 (ADX-N05, R228060, YKP10A)
12. History of phenylketonuria (PKU) or history of hypersensitivity to phenylalanine-derived products

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (59):
- United States (44):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Pulmonary Associates, Glendale, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - So Cal Institute For Respiratory Diseases, Inc., Los Angeles, California
  - Pacific Sleep Medicine, Oceanside, California
  - SDS Clinical Trials, Orange, California
  - Stanford University Center for Narcolepsy, Redwood City, California
  - Pacific Research Network, Inc., San Diego, California
  - Critical Care Pulmonary & Sleep Associates, LLC, Lakewood, Colorado
  - MD Clinical, Hallandale, Florida
  - Clinical Research Group of St. Petersburg, St. Petersburg, Florida
  - Florida Pediatric Research Institute, Winter Park, Florida
  - Emory Sleep Center, Atlanta, Georgia
  - NeuroTrials, Atlanta, Georgia
  - SleepMed of Central Georgia, Macon, Georgia
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - University of Illinois Chicago, College of Nursing, Chicago, Illinois
  - Veritas Clinical Specialties LTD, Topeka, Kansas
  - Kentucky Research Group, Louisville, Kentucky
  - The Center for Sleep & Wake Disorders, Chevy Chase, Maryland
  - Neurocare, Inc., Newton, Massachusetts
  - Clinical Neurophysiology Services, Sterling Heights, Michigan
  - Minnesota Lung Center, Edina, Minnesota
  - University of Missouri, Columbia, Missouri
  - Clayton Sleep Institute, St Louis, Missouri
  - New York University Medical center, New York, New York
  - Montefiore Medical center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Hickory Research Center, Hickory, North Carolina
  - Hickory Research Center, ARSM Research, LLC, Huntersville, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - North Coast Clinical Trials Inc., Beachwood, Ohio
  - Sleep Management Institute, Cincinnati, Ohio
  - Southwest Cleveland Sleep Research Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Sleep Medicine & Neuroscience Institute, Dublin, Ohio
  - Mercy St. Anne & Mercy St. Charles Sleep Disorders Center, Toledo, Ohio
  - Lowcountry Lung Critical Care, Charleston, South Carolina
  - Sleep Med of South Carolina, Columbia, South Carolina
  - FutureSearch Trials of Neurology LP, Austin, Texas
  - Todd J. Swick, Houston, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas
  - Swedish Medical Center, Seattle, Washington
- Canada (5):
  - London Health Sciences Centre, London, Ontario
  - Toronto Sleep Institute, Toronto, Ontario
  - Toronto Psychiatric Research Foundation, Toronto, Ontario
  - Pediatric Sleep Research Inc., Toronto, Ontario
  - CARSM Sleep Laboratory & Clinic, Montreal, Quebec
- Helsinki Sleep Clinic, Helsinki, Finland
- France (3):
  - Hospital Roger Salengro, Lille
  - Universite Paris 5 Hôtel-Dieu, Paris
  - Hopital Bichat - Claude Bernard, Paris
- Germany (5):
  - medbo Bezirksklinikum Regensburg Schlafmedizinisches Zentrum, Regensburg, Bavaria
  - Universitaetsklinikum Muenster, Münster, North Rhine-Westphalia
  - Advanced Sleep Research GmbH, Berlin
  - Studienzentrum Wilhelmshoehe, Kassel
  - Somni bene GmbH Institut für Medizinische Forschung und Schlafmedizin Schwerin GmbH, Schwerin
- Sleep Wake Center SEIN Heemstede, Heemstede, North Holland, Netherlands

REFERENCES:
- [Derived] Rosenberg R, Thorpy MJ, Dauvilliers Y, Schweitzer PK, Zammit G, Gotfried M, Bujanover S, Scheckner B, Malhotra A. Incidence and duration of common early-onset adverse events in randomized controlled trials of solriamfetol for treatment of excessive daytime sleepiness in obstructive sleep apnea and narcolepsy. J Clin Sleep Med. 2022 Jan 1;18(1):235-244. doi: 10.5664/jcsm.9550. PMID 34283019
- [Derived] Rosenberg R, Baladi M, Bron M. Clinically relevant effects of solriamfetol on excessive daytime sleepiness: a posthoc analysis of the magnitude of change in clinical trials in adults with narcolepsy or obstructive sleep apnea. J Clin Sleep Med. 2021 Apr 1;17(4):711-717. doi: 10.5664/jcsm.9006. PMID 33226332
- [Derived] Dauvilliers Y, Shapiro C, Mayer G, Lammers GJ, Emsellem H, Plazzi G, Chen D, Carter LP, Lee L, Black J, Thorpy MJ. Solriamfetol for the Treatment of Excessive Daytime Sleepiness in Participants with Narcolepsy with and without Cataplexy: Subgroup Analysis of Efficacy and Safety Data by Cataplexy Status in a Randomized Controlled Trial. CNS Drugs. 2020 Jul;34(7):773-784. doi: 10.1007/s40263-020-00744-2. PMID 32588401
- [Derived] Emsellem HA, Thorpy MJ, Lammers GJ, Shapiro CM, Mayer G, Plazzi G, Chen D, Carter LP, Villa KF, Lee L, Menno D, Black J, Dauvilliers Y. Measures of functional outcomes, work productivity, and quality of life from a randomized, phase 3 study of solriamfetol in participants with narcolepsy. Sleep Med. 2020 Mar;67:128-136. doi: 10.1016/j.sleep.2019.11.1250. Epub 2019 Dec 4. PMID 31926465

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 239 subjects were randomized in a 1:1:1:1 ratio to receive placebo, 75 mg JZP-110, 150 mg JZP-110 or 300 mg JZP-110. 236 subjects received at least 1 dose of study medication and comprised the Safety Population; the remaining 3 subjects were randomized in error (did not receive study medication) and were excluded from the Safety Population.
Groups:
- 75 mg of JZP-110: 75 mg JZP-110 administered orally, QD, for the 12-week treatment phase.
- 150 mg JZP-110: Subjects randomized to receive 150 mg JZP-110 initially received 75 mg JZP-110 from Day 1 through Day 3 of the Treatment Phase and then received 150 mg JZP-110 starting on Day 4, administered orally, QD.
- 300 mg of JZP-110: Subjects randomized to receive 300 mg JZP-110 initially received 150 mg JZP-110 from Day 1 through Day 3 of the Treatment Phase, and received 300 mg JZP-110 starting on Day 4, administered orally, QD.
- Placebo: Placebo administered orally, QD, for the 12 week treatment phase.
Period: Overall Study
Arm/Group | 75 mg of JZP-110 | 150 mg JZP-110 | 300 mg of JZP-110 | Placebo
Started | 59 | 59 | 59 | 59
Completed | 49 | 51 | 43 | 52
Not Completed | 10 | 8 | 16 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 75 mg of JZP-110 | 150 mg JZP-110 | 300 mg of JZP-110 | Placebo | Total
Number analyzed (Participants) | 59 | 59 | 59 | 59 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (12.78) | 38.1 (13.00) | 34.3 (11.51) | 36.0 (15.17) | 36.3 (12.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 42 | 40 | 35 | 154
  Male | 22 | 17 | 19 | 24 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 2
  Asian | 0 | 3 | 3 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 12 | 6 | 5 | 10 | 33
  White | 46 | 48 | 48 | 47 | 189
  More than one race | 1 | 1 | 1 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Maintenance of Wakefulness Test (MWT) From Baseline to Week 12
Description: Change in mean sleep latency time (in minutes) as determined from the first 4 trials of a 40-minute MWT from baseline to Week 12. MWT sleep latency ranges from 0 to 40 minutes, with higher scores indicating greater ability to stay awake; a positive change from baseline represents improvement in the sleep latency time. Mean sleep latency defined as the average of the first 4 MWT trials, if 3 or 4 of them are non-missing.
Time Frame: Baseline to Week 12
Population: Five subjects in the Safety Population were excluded from the mITT Population resulting in a total of 231 subjects.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | 75 mg of JZP-110 | 150 mg JZP-110 | 300 mg of JZP-110
Number analyzed (Participants) | 58 | 59 | 55 | 59
minutes | 2.12 (1.289) | 4.74 (1.335) | 9.77 (1.327) | 12.27 (1.389)

2. Primary Outcome: Change in ESS Score From Baseline to Week 12
Description: Change in Epworth Sleepiness Scale (ESS) score from Baseline to Week 12. A negative change from baseline represents improvement in excessive sleepiness.
  The ESS is a self-administered questionnaire with 8 questions. Each activity is scored on a scale ranging from 0-3, with 0 = would never fall asleep, and 3 = high chance of falling asleep. The total score ranges from 0-24, with a higher number representing an increased propensity for sleepiness. An analysis of covariance (ANCOVA) was used for the analysis of ESS scores. The response variable was the change in ESS score from baseline.
Time Frame: Baseline to Week 12
Population: Five subjects in the Safety Population were excluded from the mITT Population resulting in a total of 231 subjects.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | 75 mg of JZP-110 | 150 mg JZP-110 | 300 mg of JZP-110
Number analyzed (Participants) | 58 | 59 | 55 | 59
points on a scale | -1.6 (0.65) | -3.8 (0.67) | -5.4 (0.66) | -6.4 (0.68)

3. Secondary Outcome: Subjects Reported Improved on the Patient Global Impression of Change (PGIc) at Week 12
Description: Percentage of subjects reported as improved (minimally, much, or very much) on the PGIc at Week 12. PGIc was rated by subjects and measures the change in their condition since treatment starts on a 7-point scale ranging from 1= very much improved to 7= very much worse
Time Frame: Baseline to Week 12
Population: Five subjects in the Safety Population were excluded from the mITT Population resulting in a total of 231 subjects.
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | 75 mg of JZP-110 | 150 mg JZP-110 | 300 mg of JZP-110
Number analyzed (Participants) | 58 | 59 | 55 | 59
percentage of subjects | 39.7 | 67.8 | 78.2 | 84.7

4. Secondary Outcome: Change in Sleep Latency Time on MWT Trial 1 at Week 12
Description: Time course of efficacy in MWT: Change in sleep latency (in minutes) on each of the 5 MWT trials at Week 12.
Time Frame: Change from baseline for sleep latency in MWT during trial 1 at week 12
Population: Five subjects in the Safety Population were excluded from the mITT Population resulting in a total of 231 subjects.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | 75 mg of JZP-110 | 150 mg JZP-110 | 300 mg of JZP-110
Number analyzed (Participants) | 58 | 59 | 55 | 59
minutes | -0.55 (4.658) | 3.27 (1.725) | 9.87 (1.713) | 9.91 (1.841)

5. Secondary Outcome: Change in Sleep Latency Time on MWT Trial 2 at Week 12
Description: Time course of efficacy in MWT: Change in sleep latency (in minutes) on each of the 5 MWT trials at Week 12.
Time Frame: Change from baseline for sleep latency in MWT during trial 2 at week 12
Population: Five subjects in the Safety Population were excluded from the mITT Population resulting in a total of 231 subjects.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | 75 mg of JZP-110 | 150 mg JZP-110 | 300 mg of JZP-110
Number analyzed (Participants) | 58 | 59 | 55 | 59
minutes | 1.41 (1.638) | 5.70 (1.697) | 9.46 (1.674) | 14.50 (1.835)

6. Secondary Outcome: Change in Sleep Latency Time on MWT Trial 3 at Week 12
Description: Time course of efficacy in MWT: Change in sleep latency (in minutes) on each of the 5 MWT trials at Week 12.
Time Frame: Change from baseline for sleep latency in MWT during trial 3 at week 12
Population: Five subjects in the Safety Population were excluded from the mITT Population resulting in a total of 231 subjects.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | 75 mg of JZP-110 | 150 mg JZP-110 | 300 mg of JZP-110
Number analyzed (Participants) | 58 | 59 | 55 | 59
minutes | 3.79 (1.799) | 6.35 (1.908) | 11.31 (1.859) | 13.99 (1.996)

7. Secondary Outcome: Change in Sleep Latency Time on MWT Trial 4 at Week 12
Description: Time course of efficacy in MWT: Change in sleep latency (in minutes) on each of the 5 MWT trials at Week 12.
Time Frame: Change from baseline for sleep latency in MWT during trial 4 at week 12
Population: Five subjects in the Safety Population were excluded from the mITT Population resulting in a total of 231 subjects.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | 75 mg of JZP-110 | 150 mg JZP-110 | 300 mg of JZP-110
Number analyzed (Participants) | 58 | 59 | 55 | 59
minutes | 2.33 (1.579) | 3.77 (1.663) | 9.77 (1.606) | 13.50 (1.734)

8. Secondary Outcome: Change in Sleep Latency Time on MWT Trial 5 at Week 12
Description: Time course of efficacy in MWT: Change in sleep latency (in minutes) on each of the 5 MWT trials at Week 12.
Time Frame: Change from baseline for sleep latency in MWT during trial 5 at week 12
Population: Five subjects in the Safety Population were excluded from the mITT Population resulting in a total of 231 subjects.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | 75 mg of JZP-110 | 150 mg JZP-110 | 300 mg of JZP-110
Number analyzed (Participants) | 58 | 59 | 55 | 59
minutes | 3.09 (1.808) | 3.92 (1.928) | 9.25 (1.888) | 12.20 (1.969)

9. Secondary Outcome: Change in the Mean Sleep Latency Time as Determined From the First 4 Trials of a 40-Minute MWT From Baseline to Week 4
Description: Change in mean sleep latency time (in minutes) as determined from the first 4 trials of a 40-minute MWT from Baseline to Week 4.
Time Frame: Baseline to Week 4
Population: Five subjects in the Safety Population were excluded from the mITT Population resulting in a total of 231 subjects.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | 75 mg of JZP-110 | 150 mg JZP-110 | 300 mg of JZP-110
Number analyzed (Participants) | 58 | 59 | 55 | 59
minutes | 2.16 (1.202) | 4.67 (1.223) | 9.15 (1.246) | 13.07 (1.211)

ADVERSE EVENTS:
Time Frame: Through Week 14
Arm/Group | Placebo | 75 mg of JZP-110 | 150 mg JZP-110 | 300 mg of JZP-110
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59 | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59 | 1/59 | 0/59
Other Adverse Events (participants affected / at risk) | 17/59 | 19/59 | 32/59 | 36/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=59) | 75 mg of JZP-110 (N=59) | 150 mg JZP-110 (N=59) | 300 mg of JZP-110 (N=59)
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=59) | 75 mg of JZP-110 (N=59) | 150 mg JZP-110 (N=59) | 300 mg of JZP-110 (N=59)
Weight decreased (Investigations) | 0 | 1 | 1 | 3
Heart rate increased (Investigations) | 0 | 0 | 0 | 4
Weight increased (Investigations) | 3 | 2 | 0 | 1
Headache (Nervous system disorders) | 3 | 6 | 14 | 18
Dizziness (Nervous system disorders) | 2 | 2 | 1 | 3
Fatigue (General disorders) | 0 | 0 | 2 | 3
Anxiety (Psychiatric disorders) | 1 | 1 | 3 | 5
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 3
Nausea (Gastrointestinal disorders) | 1 | 3 | 6 | 6
Dry mouth (Gastrointestinal disorders) | 2 | 3 | 4 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2 | 3
Constipation (Gastrointestinal disorders) | 1 | 3 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 5 | 5 | 9
Nasopharyngitis (Infections and infestations) | 3 | 5 | 8 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 4 | 0
Influenza (Infections and infestations) | 3 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review trial results communications prior to public release and can embargo such communications for a period of at least 60 days from the time submitted to sponsor for review. If requested by sponsor, the PI will withhold publication for up to an additional 30 days. Furthermore, the first publication of study results must be a joint publication of all study sites unless a joint manuscript has not been submitted for publication within 12 months of completion of the study.

DOCUMENTS (2):
  • Study Protocol (2016-02-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT02348593/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT02348593/SAP_001.pdf